CLINICAL TRIAL: NCT03445624
Title: Abdominal Ultrasound With Doppler and Peripheral Hemogram in Assesment Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hyam fathy, clinical professor, Assiut University
Other Study IDs: assiut hospitals university
Record Dates: First submitted 2018-01-09; First posted 2018-02-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab; Steroids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patient on traditional therapy: Drug: steroid,5ASA , immuran for assesment the outcome of therapy in inflammatory bowel disease steroid(40- 60mg tablet),5ASA(pentasa 3-4gm tablet),azathioprin (immuran 100 mg tablet)
  Interventions: Drug: Infliximab
- patient on infliximab: drug : infliximab (5mglkg intravenous)for the first dose,the second dose after 2 weeks the third dose after 6 weeks then every 2 months
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — follow up the patients who received this drugs for 1 year by abdominal ultrasound,peripheral hemogram and colonoscopy
  Other Names: steroid,immuran 5ASA

SUMMARY:
assessment of inflammatory bowel disease patients in activity and remission by abdominal ultrasound examine non-invasive and in physiological condition by measuring the colon wall thickness in diagnosis and follow up the patient also including extra intestinal features such as the splanchnic vessels,mesentery and lymph nodes . Doppler u.s can evaluate bowel wall vascularity In activity and remission . peripheral hemogram in relationship to activity inflammatory bowel disease asses anemia ,increase monocyte and decrease mean platelet volume( MPV) . also,the investigator will evaluate the outcome of different lines of treatment traditional and biologic therapy (response to treatment,times of activity and complications)

DETAILED DESCRIPTION:
the participants will follow up the patient for 1 year in the first visit

All patients in this study will be subjected to:

1. Detailed history.
2. Careful physical examination
3. laboratory investigation

   1. complete blood picture.
   2. liver function
   3. kidney function
   4. Iron profile(serum iron ,serum ferritin
   5. ESR (erythrocyte sedimentation rate )

   g-CRP (C reactive protein) f-LDH (lactate dehydrogenase)
4. Abdominal us(the colon wall thickness,lymph nodes,mass,other organs)
5. Doppler us (mesenteric vessels)
6. colonoscopy after 1 year of treatment follow up every 3 months by abdominal US and peripheral hemogram and last visit after 1 year colonoscopy and biopsy for assessment response to treatment

ELIGIBILITY:
Inclusion Criteria

* patients diagnosed ulcerative colitis at age(15-60)
* patients diagnosed crohns disease at age(15-60)k

Exclusion criteria

* liver cirrhosis and portal hypertension
* spontaneous bacterial peritonitis
* Ischemic colitis

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patients diagnosed inflammatory bowel disease (ulcerative colitis and crohns disease) at age(15 -60)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
the role abdominal ultrasound in assessment inflammatory bowel disease | 2 year
  measure the thickness of the colon by abdominal ultrasound and doppler mesenteric vessels .more than 4ml detect activity doppler mesenteric highly vascularity in activity

OTHER OUTCOMES:
Assesment inflammatory bowel disease by complete blood picture | 2year
  follow up haemoglobin level (less than 10 mg) indicate anemia which mean the patient uncontrolled monocyte( monocyte more than 12% of white blood cell count detect activity) Mean platelet volume less than 6 fl which decrease in activity inflammatory bowel disease

CONTACTS AND LOCATIONS:
Overall Officials: ahmed ashmawy, Study Director — lecturer of internal medicine
Locations (1):
- Hyam Fathy, Asyut, Egypt